CLINICAL TRIAL: NCT02106416
Title: Development of a Novel Technique for PET/MRI Tracer Kinetic Analysis for Urologic Pelvic Malignancy
Brief Title: Use of PET/MRI Tracer to Further Understanding of Prostate Cancer Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-00394
Record Dates: First submitted 2013-10-25; First posted 2014-04-08 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer; Bladder Cancer
Keywords: prostate cancer; bladder cancer; MRI; PET; perfusion
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/MRI (Experimental): Patient receives PET/MRI
  Interventions: Procedure: PET/MRI

INTERVENTIONS:
Procedure: PET/MRI — Simultaneous PET/MRI (3T system)
  Other Names: Siemens Biograph mMR

SUMMARY:
The purpose of this study is to develop a novel technique for integrated PET/MRI tracer kinetic analysis for urologic malignancy.

DETAILED DESCRIPTION:
Patients scheduled to undergo gadolinium-enhanced MRI for urologic malignancy will be recruited to undergo PET/MRI employing simultaneous dynamic acquisition of PET and gadolinium-chelate data sets. For initial technical development within this pilot study, analysis will be performed attempting to compute tracer delivery using inputs from an integrated MRI-perfusion analysis. Flow and permeability will be obtained from the MR perfusion analysis, which can be used to compute the inflow rate constant K1. K1, reflecting the transfer of contrast, will then be used to compute the metabolic uptake of FDG by the organ as well as of any visible tumors. A determination will be made whether this metabolic uptake is successfully computed for each case. If not, then acquisition and post-processing modifications will be made for subsequent cases.

ELIGIBILITY:
Inclusion Criteria:

The study population will consist of patients with known urologic cancer who are scheduled to undergo MRI with gadolinium for their routine care. Patients will be referred by the Urology or Medical Oncology Departments for participation in the study. Subjects will be selected on the basis of their willingness and ability to participate and on their likelihood of completing the study. Patients agreeing to participate will be presented with a flyer which will inform subject about the available research study and study contact information. participation is entirely voluntary, and a subject may withdraw from the study at any time. Normal volunteers will be recruited accessing the existing database of normal volunteers maintained in Radiology Research department.

Exclusion Criteria:

Normal MRI exclusion criteria will apply, including those on the following list. A standard MRI safety form will be used to identify potential conditions warranting exclusion.

* Electrical implants such as cardiac pacemakers or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial heart, valves with steel parts, metal fragments, shrapnel, bullets, tattoos near the eye, or steel implants
* Ferromagnetic objects such as jewelry or metal clips in clothing
* Claustrophobia
* History of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The inflow rate constant K1 | Within six months of scan completion
  The inflow rate constant K1 will be calculated based on assessment of dynamic PET/MRI data.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rosenkrantz, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States